CLINICAL TRIAL: NCT01610167
Title: NUPRO(r) Sensodyne Prophylaxis Paste With NovaMin(r) for the Treatment of Dentin Hypersensitivity.
Brief Title: NUPRO(r) Sensodyne Prophylaxis Paste With NovaMin(r)Sensitivity Relief Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-001
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Tooth Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NUPRO(r) Classic Prophy Paste (Active Comparator)
  Interventions: Device: NUPRO Classic Prophy Paste
- NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ fluoride. (Experimental)
  Interventions: Device: NUPRO Sensodyne Prophy Paste with Novamin with fluoride.
- NUPRO Sensodyne Prophy Paste w/ Novamin (Experimental)
  Interventions: Device: NUPRO Sensodyne Prophy Paste with Novamin without fluoride.

INTERVENTIONS:
Device: NUPRO Classic Prophy Paste — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Arms: NUPRO(r) Classic Prophy Paste
Device: NUPRO Sensodyne Prophy Paste with Novamin with fluoride. — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Arms: NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ fluoride.
Device: NUPRO Sensodyne Prophy Paste with Novamin without fluoride. — Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
  Arms: NUPRO Sensodyne Prophy Paste w/ Novamin

SUMMARY:
The study is intended to verify through clinical measurement that the NUPRO Sensodyne Prophylaxis Paste with Novamin provides immediate sensitivity relief as well as extended relief up to 28 days.

DETAILED DESCRIPTION:
It is hypothesized that the prophy paste with NovaMin(r)will give patients immediate sensitivity relief, as well as sensitivity relief up to 4 weeks (28 days) after measurement.

ELIGIBILITY:
Inclusion Criteria:

* Availability to complete in the 28 day duration of the study.
* Two sensitive teeth which are not adjacent to each other and preferably in different quadrants and demonstrate cervical erosion, abrasion, and gingival recession.
* qualifying response to tactile stimuli as defined by a score of </= 20 grams.
* Qualifying response to air blast stimuli as defined by a score of >/= 1 on the Schiff Cold Air Sensitivity Scale.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for 3 weeks prior to entry into the study.
* Able to follow study procedures and instructions.
* Must have a minimum of 10 natural evaluable teeth, excluding 3rd molars.

Exclusion Criteria:

* Individuals who exhibit gross oral pathology
* Females who may be pregnant or lactating or intending to become pregnant
* Individuals who require anesthetic during scaling
* Dental pathology which may cause pain similar to tooth sensitivity
* Individuals with large amounts of calculus
* Subjects with active infectious diseases such as hepatitis, HIV or tuberculosis
* Any condition requiring antibiotic prophylaxis for dental treatment
* Excessive gingival inflammation
* Individuals who had their teeth cleaned within 30 days of the screening appointment
* Individuals who have had a desensitizing treatment or tooth bleaching within 90 days of screening appointment.
* Oral pathology, chronic disease, or history of allergy to test products
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Regular use of sedatives, anti-inflammatory drugs, or analgesic
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past 4 weeks.
* Current participation in any other clinical study or receipt of an investigational drug within 30 days of the screening visit at the start of the study.
* Personnel; a) An employee of the sponsor; b) A member or relative of the study site staff directly involved with the study.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Any subject who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L. Milleman, DDS, MPA, Principal Investigator — Salus Research; Kimberly R. Milleman, ASDH, MS, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 327 subjects queried from Investigator database following IRB apprvoal on 14-Sept.-2011. 199 of the queried subjects were consented and screened. 161 subjects were accepted at screening and appointed for baseline visit 2 weeks later. 159 subjects were evaluated at the baseline exam and 151 subjects were randomized and enrolled into the study.
Pre-assignment Details: 10 subjects were lost following screening and at baseline assessment. 5 of the 10 were disqualified due to insufficient tactile response, 3 due to lack of evaproative hypersensitivity, and 2 had scheduling conflicts.
Groups:
- NUPRO Sensodyne Prophy Paste w/ Novamin: NUPRO Sensodyne Prophy Paste with Novamin without fluoride. : Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
- NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride.: NUPRO Sensodyne Prophy Paste with Novamin with fluoride. : Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
- NUPRO(r) Classic Prophy Paste: NUPRO Classic Prophy Paste : Abrasive, flavored dental prophylaxis paste for cleaning and polishing teeth.
Period: Overall Study
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Started | 52 | 49 | 50
Completed | 52 | 49 | 48
Not Completed | 0 | 0 | 2
Not completed — Scheduling conflict. | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste | Total
Number analyzed (Participants) | 52 | 49 | 50 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 52 | 49 | 49 | 150
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.31 (11.10) | 41.55 (10.70) | 42.10 (10.31) | 41.65 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 35 | 107
  Male | 15 | 14 | 15 | 44
Region of Enrollment [Number; unit: participants]
  United States | 52 | 49 | 50 | 151

OUTCOME MEASURES:

1. Primary Outcome: Immediate Sensitivity Relief. Tactile Sensitivity.
Description: Assessment of sensitivity via tactile stimulation immediately after treatment. Tactile sensitivity measured using a Yeaple probe recording tactile pressure in grams before nerve stimulation. Point of nerve stimulation identified by patient with a "yes" response as pressure is increased in 10 gram increments. Tactile sensitivity is reported as the change from baseline after treatment.
Time Frame: Immediately after treatment.
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Number analyzed (Participants) | 52 | 49 | 50
grams | 12.36 (12.91) | 10.46 (12.58) | 0.60 (3.45)

2. Primary Outcome: Adverse Events.
Description: Assessment of adverse events that may occur as a result of treatment (typically includes any kind of allergic reation to paste).
Time Frame: Immediately after treatment to 28 days (+/- 2 days) post treatment.
Population: Intent to treat (ITT).
Measure: Number; unit: Number of adverse events.
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Number analyzed (Participants) | 52 | 49 | 50
Number of adverse events. | 0 | 0 | 0

3. Secondary Outcome: Extended Sensitivity Relief. Tactile Sensitivity.
Description: Assessment of sensitivity score via tactile stimulation 28 days post treatment. Tactile sensitivity measured using a Yeaple probe recording tactile pressure in grams before nerve stimulation. Point of nerve stimulation identified by patient with "yes" response as pressure is increased in 10 gram increments. Measured sensitivity is reported as difference from baseline examination.
Time Frame: 28 days (+/- 2 days) post treatment.
Population: Intent to treat (ITT).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Number analyzed (Participants) | 52 | 49 | 48
grams | 10.19 (11.37) | 11.07 (11.90) | 1.15 (5.88)

4. Primary Outcome: Immediate Sensitivity Relief. Air Blast Sensitivity.
Description: Sensitivity measurements performed using a cold air blast and sensitivity scored on the four (4) point Schiff scale with 0 equal to no discomfort or awareness of sensitivity and 3 equal to severe pain from sensitive teeth. Score is reported as the change from baseline after treatment.
Time Frame: Immediately after treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Number analyzed (Participants) | 52 | 49 | 50
units on a scale | -0.87 (0.71) | -0.86 (0.62) | 0.00 (0.35)

5. Secondary Outcome: Extended Sensitivity Relief. Air Blast Sensitivity.
Description: Assessment of cold air sensitivity. Cold air sensitivity measurements performed using a cold air blast and sensitivity scored on the four (4) point Schiff scale with 0 equal to no discomfort or awareness of sensitivity and 3 equal to severe pain from sensitive teeth.
Time Frame: 28 days (+/- 2 days) post treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Number analyzed (Participants) | 52 | 49 | 48
units on a scale | -0.94 (0.68) | -0.95 (0.66) | 0.03 (0.47)

ADVERSE EVENTS:
Arm/Group | NUPRO Sensodyne Prophy Paste w/ Novamin | NUPRO Sensodyne Prophy Paste w/ Novamin(r) w/ Fluoride. | NUPRO(r) Classic Prophy Paste
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less